CLINICAL TRIAL: NCT00267423
Title: A Single Center, Retrospective Study of the Safety and Feasibility of Epicardial Biventricular Pacing in the Pediatric Population
Brief Title: Biventricular Pacing in the Pediatric Population
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 04-040
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; electrophysiology; epicardial biventricular pacing
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Hypothesis 1 (H1): Epicardial biventricular pacing is a safe and feasible method of pacing in young patients.

Over the last two years, physicians at Children's Healthcare of Atlanta have been implanting epicardial BiV pacing systems in children determined to have ventricular dyssynchrony caused by numerous cardiac diagnoses. The decision to use these pacing systems was based on the knowledge gained by adult studies. Since the use of these pacing systems in the pediatric population has not been formally studied, we propose a study to retrospectively review the safety and feasibility of epicardial BiV pacing in pediatric patients. This study will involve the review of the medical records of children who received epicardial BiV systems at Children's Healthcare of Atlanta between January 2002 and May 2004.

DETAILED DESCRIPTION:
Synchronous activation of the right and left ventricles requires a normally functioning sinoatrial (SA) node, atrioventricular (AV) node and ventricular conduction system. When AV conduction has been interrupted by congenital heart block or acquired damage to the AV node, impulses arising from the SA node do not reach the ventricular myocardium. Standard therapy involves the placement of a permanent pacing system. In young children, such a system consists of either placing a single epicardial pacing lead on the right ventricular (RV) surface or separate epicardial pacing leads placed on the right atrium (RA) and RV. The former is commonly referred to as single chamber pacing and the latter as dual chamber pacing [AV sequential, single-site (SS) ventricular pacing]. The decision regarding single versus dual chamber lead placement is heavily influenced by operator convenience in the setting of a limited sternotomy. The main functions of the pacing system are sensing spontaneous activity and delivering pacing stimuli when appropriate. The two major advantages of dual chamber pacing are maintenance of physiologic heart rates and restoration of AV synchrony. The disadvantage of this system, however, is that the intrinsic synchronous depolarization of the ventricles is interrupted by initial paced ventricular activation in the RV rather than via the specialized His-Purkinje system; thus desynchronizing ventricular electrical activation. In addition, recent studies have demonstrated that despite early institution of cardiac pacing, some infants and children with AV block (AVB) develop late-onset left ventricular (LV) dilated cardiomyopathy over a follow-up period of 10 years.(1) The underlying mechanisms for this cardiomyopathy are not clear. A novel method of pacing (biventricular pacing, BiV) has been used in adult patients with left bundle branch block (LBBB, which results in dysynchronous ventricular activation) and congestive heart failure (CHF). Biventricular pacing in adults involves transvenous endocardial pacing leads placed in the RA, RV apex and LV via the coronary sinus. This results in "resynchronization" of ventricular activation, presumably by restoring a "normal" ventricular activation sequence, and has been associated with decreased CHF symptoms and improved ventricular function.

Children with acquired or congenital AVB, on the other hand, typically have a narrow QRS; owing to a midline ventricular escape rhythm and synchronous ventricular activation. The typical modes of pacing (VVI or DDD, single-site ventricular) in these children result in interventricular dyssynchrony, as described above. Recent studies in adult populations (DAVID, AAIR vs. DDDR in SSS, and MOde Selection trials)(2-4) demonstrated the detrimental effects of standard single-site ventricular pacing. Unfortunately, children with acquired and/or congenital AVB do not have the option of pacing or no pacing, and are destined to potentially decades of being 100% ventricular paced. This further emphasizes the importance of optimizing pacing strategies in this young, vulnerable population.

Specific Aim 1 (SA1): To evaluate the safety and feasibility of biventricular epicardial pacing in children.

ELIGIBILITY:
Inclusion Criteria:

* any pediatric patient who received an epicardial BiV pacing system at Children's Healthcare of Atlanta between January 2002 and May 2004.

Exclusion Criteria:

* those patients who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Frias, MD, Principal Investigator — Sibley Heart Center Cardiology at Children't Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States